CLINICAL TRIAL: NCT03805789
Title: A Phase 2/3, Multicenter, randOmized, Double-blind, Placebo-controlled, stUdy to evaLuate the Safety and Efficacy of Alpha-1 AntiTrypsin for the prEvention of Graft-versus-host Disease in Patients Receiving Hematopoietic Cell Transplant (MODULAATE Study)
Brief Title: The Safety and Efficacy of Alpha-1 Antitrypsin (AAT) for the Prevention of Graft-versus-host Disease (GVHD) in Patients Receiving Hematopoietic Cell Transplant
Acronym: MODULAATE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL964_2001; 2018-000329-29 (EudraCT Number); 2024-511164-92-00 (EU CTIS Number)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Acute-graft-versus-host Disease
MeSH Terms: interventions — alpha 1-Antitrypsin; Respreeza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AAT (low dose) (Experimental): Open label. AAT is a lyophilized product for intravenous (IV) administration
  Interventions: Biological: AAT
- AAT (medium dose) (Experimental): Open label. AAT is a lyophilized product for IV administration
  Interventions: Biological: AAT
- AAT (high dose) (Experimental): Open label. AAT is a lyophilized product for IV administration
  Interventions: Biological: AAT
- AAT (selected dose from open-label) (Experimental): Double-blind. AAT is a lyophilized product for IV administration
  Interventions: Biological: AAT
- Placebo (Placebo Comparator): Albumin solution administered intravenously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AAT — AAT is a lyophilized product for IV administration.
  Other Names: Alpha-1 proteinase inhibitor; Respreeza
  Arms: AAT (high dose); AAT (low dose); AAT (medium dose); AAT (selected dose from open-label)
Biological: Placebo — Albumin solution administered intravenously
  Arms: Placebo

SUMMARY:
This study is a phase 2 / 3 prospective, double-blind, randomized, multicenter, placebo-controlled study for prevention of acute GVHD (aGVHD) in participants undergoing an unrelated (matched or single allele mismatched) or matched related allogeneic hematopoietic cell transplantation (HCT).

ELIGIBILITY:
Inclusion Criteria:

* • Male or female participants, >=12 years of age (>= 18 years of age for participants at German sites only), undergoing HCT for hematological malignancies, including leukemia, lymphoma, multiple myeloma, myelodysplastic syndrome, and myeloproliferative neoplasms.
* • Planned myeloablative conditioning regimen.
* • Participants must have a related or unrelated donor as follows:
* - Related donor must be a 6 / 6 match for human leukocyte antigen (HLA)-A, -B, at intermediate (or higher) resolution, and -DR beta 1 (DRB1) at high resolution using deoxyribonucleic acid (DNA)-based typing.
* - Unrelated donor must be 7 / 8 or 8 / 8 match for HLA-A, -B, and -C at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing.

Exclusion Criteria:

* • Prior autologous or allogeneic HCT.
* • T cell depleted transplant or planned use of anti-T cell antibody therapy either ex vivo or in vivo (ie, anti thymocyte globulin [ATG], alemtuzumab) for GVHD prophylaxis.
* • Planned umbilical cord blood transplant.
* • Planned use of cyclophosphamide after HCT for GVHD prophylaxis.
* • Planned haploidentical donor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The time to Grade II-IV aGVHD or death | Through 180 days after HCT
  Acute GVHD will be assessed using the Harris scoring system.

SECONDARY OUTCOMES:
Proportion of participants with lower gastrointestinal (GI) aGVHD or Grade III-IV aGVHD in any organ | Through 180 days after HCT
Proportion of participants with severe infections defined by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) greater than or equal to (>=) Grade 3 | Through Day 60 after HCT
Proportion of participants with Grade II-IV aGVHD or death | Through 100 days and 180 days after HCT
Proportion of participants with lower GI aGVHD | Through Days 60, 100 and 180 after HCT
Proportion of participants with severe infections defined by NCI-CTCAE >= Grade 3 | Through 100 and 180 days after HCT
Number of deaths (relapse and nonrelapse-related) | Within 180, 365, and 730 days after HCT
  Death by any cause
Proportion of participants with Grade III-IV aGVHD or death | Through Days 60, 100, and 180 days after HCT
Proportion of participants with moderate to severe chronic GVHD | Within 180, 365, 545, and 730 days after HCT
  Moderate to severe chronic GVHD graded according to National Institutes of Health (NIH) scale.
Proportion of participants who have discontinued immune suppression therapies including standard of care GVHD prophylaxis and steroid treatment | Within 180 and 365 days after HCT
Time to neutrophil engraftment | Through 365 days after HCT
  Time to the first of 3 consecutive days of absolute neutrophil counts ≥ 500/µL.
Time to GVHD relapse-free survival | Within 365 and 730 days after HCT
  GVHD free, relapse free, survival defined as time to any of the following events: 1) Grade III-IV acute GVHD, 2) moderate-severe chronic GVHD, 3) primary malignancy relapse or 4) death.
Proportion of participants with relapse of primary malignancies | Through 180, 365, and 730 days after HCT
Proportion of participants with Grade II-IV aGVHD with an overall (complete + partial) response, complete response and partial response | Approximately 4 weeks after the initiation of systemic steroids during 8-week Treatment Period
Percent of participants with study drug related adverse events | Up to 365 days after HCT
Maximum concentration (Cmax) of AAT | Before and up to 72 after infusion of AAT
Area under the concentration curve (AUC) for AAT | Before and up to 72 after infusion of AAT
Ctrough of AAT | Before and up to 72 after infusion of AAT
Clearance (CL) of AAT | Before and up to 72 after infusion of AAT
Volume of distribution (V) for AAT | Before and up to 72 after infusion of AAT

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — CSL Behring
Locations (34):
- United States (12):
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Johns Hopkins Hospital, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - The University of Texas-MD Anderson Cancer Center, San Antonio, Texas
  - University of Utah Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Royal Brisbane and Women's Hospital, Herston, Queenland, Australia
- Uniklinik Köln, Cologne, Germany
- Italy (2):
  - University Hospital Catania, Calabria, Catania
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Calabria
- Japan (9):
  - Anjo Kosei Hospital, Anjo-shi
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - Hiroshima University Kasumi Campus, Hiroshima
  - Aichi Medical Center Nagoya Daiichi Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
- South Korea (4):
  - INJE University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Universitario Valle de Hebron, Barcelona
  - Marqués de Valdecilla University Hospital, Barcelona
  - Salamanca University Hospital, Salamanca
- Turkey (Türkiye) (2):
  - Ankara Abdurrahman Yurtaslan, Ankara
  - Turgut Ozal Medicine Center, Battalgazi

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.